CLINICAL TRIAL: NCT07075120
Title: Pilot Study of Ipilimumab and Nivolumab With Response-adapted Stereotactic Body Radiotherapy Followed by Definitive Resection for Patients With Locally Advanced Hepatocellular Cancer
Brief Title: Ipilimumab and Nivolumab With SBRT in Locally Advanced Hepatocellular Cancer
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Hawaii (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACOBA-2024-1
Record Dates: First submitted 2025-06-20; First posted 2025-07-20 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Hepatocellular Carcinoma (HCC)
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Ipilimumab; Nivolumab; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ipilimumab and Nivolumab with SBRT and Surgical Resection (Experimental): Arm A: Patients receive ipilimumab 3mg/kg and nivolumab 1mg/kg for nine weeks (three cycles). Following completion of preoperative immunotherapy, imaging with CT or MRI is performed to determine resectability. Eligible patients proceed to surgical resection.
  Arm B: Patients who are not eligible for resection continue immunotherapy (ipilimumab and nivolumab) for one additional cycle, then nivolumab 480mg every four weeks combined with stereotactic body radiotherapy (SBRT). SBRT is administered in 3-5 fractions, and patients continue imaging every nine weeks. Surgical resection is performed once resectability is confirmed.
  Interventions: Drug: Ipilimumab and Nivolumab; Radiation: Stereotactic Body Radiotherapy (SBRT)

INTERVENTIONS:
Drug: Ipilimumab and Nivolumab — Immunotherapy combination (Ipilimumab and Nivolumab) targeting CTLA-4 and PD-1 pathways to enhance immune response.
Radiation: Stereotactic Body Radiotherapy (SBRT) — High-dose radiation therapy delivered in 3-5 fractions for local control of tumors in combination with immunotherapy. Radiation dosages are based on the RTOG 1112 trial guidelines to minimize normal tissue exposure.

SUMMARY:
Hepatocellular carcinoma (HCC) is a major cause of cancer-related deaths globally, with Native Hawaiian and Pacific Islander (NHPI) populations experiencing significantly higher mortality rates compared to other groups in Hawaii. This disparity is influenced by factors such as higher prevalence of chronic hepatitis B, non-alcoholic fatty liver disease, limited access to early detection, and delayed diagnoses. NHPI patients are also underrepresented in clinical trials, limiting the relevance of treatment advances for this population.

The standard treatment for HCC is surgical resection; however, many NHPI patients present with unresectable disease. Recent advances with immune checkpoint inhibitors (ICIs), such as nivolumab and ipilimumab, have shown promise in treating advanced HCC and improving survival in previously untreatable cases. Additionally, stereotactic body radiotherapy (SBRT) has been shown to enhance survival and local control when combined with systemic therapies like ICIs. However, without surgery, outcomes remain suboptimal, with response rates for ICIs alone at 20-30%, and combination ICI-SBRT treatment showing slightly better results but still a high risk of progression.

Despite improvements in HCC treatment, significant gaps remain in managing borderline resectable disease, especially in NHPI patients. This study aims to evaluate the safety and efficacy of combining ICIs and SBRT with curative surgery for patients with borderline resectable HCC, focusing on NHPI populations. The study will also explore the use of biomarkers such as cell-free DNA (cfDNA), CD8+ T-cell infiltration, and serum cytokine markers to guide personalized treatment strategies. Preliminary findings suggest that this multimodal approach may improve outcomes and enable surgical resection for patients previously considered inoperable.

This study seeks to address the unmet need for effective treatment strategies in borderline resectable HCC and to improve survival outcomes for underserved NHPI populations.

ELIGIBILITY:
Main Criteria for Inclusion/Exclusion

* Inclusion Criteria:

  * Histologically or cytologically confirmed hepatocellular cancer
  * Locally advanced/borderline resectable HCC as defined by:

    * Solitary tumor >5 cm, OR
    * Unilobar multifocal disease either with >3 tumors or one tumor >3 cm, OR
    * Bilobar disease with adequate future liver remnant, still technically resectable, OR
    * High risk disease features (tumor >3 cm with macrovascular invasion or tumor >3 cm with AFP>400).
  * No extrahepatic spread, no nodal disease, no bilateral left and right branch portal vein involvement, no hepatic vein / IVC involvement. Unilateral hepatic vein involvement is not exclusionary.
  * Measurable disease per RECIST 1.1 as determined by the investigator
  * Age ≥ 18 years old on the day of consent
  * ECOG performance status ≤1 (Appendix XX)
  * Adequate organ and marrow function, as defined below. Criteria "a," "b," "c," and "f" cannot be met with transfusions, infusions, or growth factor support administered within 14 days of starting the first dose.

    * Hemoglobin ≥9 g/dL
    * Absolute neutrophil count ≥1000/μL
    * Platelet count ≥90,000/μL
    * Total bilirubin (TBL) <2.0 mg/dL
    * ASTandALT≤5×ULN
    * Albumin≥2.8g/dL
    * International normalized ratio(INR)≤2xULN
    * Calculated creatinine clearance ≥ 40 mL/minute as determined by Cockcroft-Gault (using actual body weight) or 24-hour urine creatinine clearance
* Exclusion Criteria:

  * Prior systemic therapy for hepatocellular carcinoma
  * Radiotherapy treatment to more than 30% of the bone marrow or with a wide field of radiation within 28 days of the first dose of study drug(s).
  * Ascites that requires ongoing paracentesis, within 6 weeks prior to the first scheduled dose, to control symptoms.
  * Active or prior documented GI variceal bleed or history of upper GI bleeding, ulcers, or esophageal varices with bleeding within 60 days prior to registration; adequate endoscopic therapy according to institutional standards is required for patients with history of esophageal variceal bleeding or assessed as high risk for esophageal variceal by the treating investigator.
  * Hepatic encephalopathy within 12 months of trial registration
  * Patient currently exhibits symptomatic or uncontrolled hypertension defined as diastolic blood pressure >90 mmHg or systolic blood pressure >140 mmHg.
  * Prior external beam radiation therapy to the liver, prior yttrium-90 radioembolization
  * HBV viral load >100 IU/mL, ongoing corticosteroid therapy >10 mg prednisone daily, and active autoimmune disease requiring systemic therapy in the past 2 years.
  * Direct tumor extension into stomach, duodenum, small or large bowel
  * Active or untreated central nervous system (CNS) and leptomeningeal metastases
  * History of another primary malignancy except for:

    * Malignancy treated with curative intentand with no known active disease ≥ 5years before the first dose of study drug(s) and of low potential risk for recurrence
    * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
    * Adequately treated carcinoma in situ without evidence of disease
  * Known fibrolamellar HCC, sarcomatoid HCC, or mixed cholangiocarcinoma and HCC.
  * Active infection including tuberculosis (TB) (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice), or human immunodeficiency virus (positive human HIV 1/2 antibodies).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Treatment Regimen | From treatment initiation to surgery completion (up to 12 months)
  Feasibility will be defined as fewer than 5 failures of resection due to treatment-related factors (e.g., toxicity, delay in treatment).
  (Co-primary endpoint; this outcome assesses the tolerability and logistical feasibility of the neoadjuvant treatment strategy.) Unit of Measure: Number of failures (count)
R0 Resection Rate | From treatment initiation to surgery (up to 12 weeks)
  The proportion of patients achieving R0 surgical resection, defined as complete resection with negative margins.
  (Co-primary endpoint; this outcome reflects the treatment's impact on surgical resectability.) Unit of Measure: Percentage of participants

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | From the date of treatment initiation until the date of best documented response, assessed up to 36 months.
  ORR will be assessed based on RECIST v1.1 criteria.
Pathologic Complete Response (pCR) and Disease-Free Survival (DFS) | From the date of treatment initiation until disease recurrence or progression, assessed up to 36 months.
  pCR and DFS will be evaluated as secondary endpoints.
Overall Survival (OS) | From the date of treatment initiation until death, assessed up to 36 months.
  OS will be estimated from the date of treatment initiation to the date of death.
Toxicity Evaluation | From the start of treatment to the time of surgery, assessed up to 12 months.
  Toxicity will be evaluated using the CTCAE v6.0 grading system for grade 3-4 adverse events prior to surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Jared D Acoba, MD, Principal Investigator — University of Hawaii
Locations (1):
- University of Hawai'i Cancer Center, Honolulu, Hawaii, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chopra S, George K, Engineer R, Rajamanickam K, Nojin S, Joshi K, Swamidas J, Shetty N, Patkar S, Patil P, Ostwal V, Mehta S, Goel M. Stereotactic body radio therapy for inoperable large hepatocellular cancers: results from a clinical audit. Br J Radiol. 2019 Sep;92(1101):20181053. doi: 10.1259/bjr.20181053. Epub 2019 Jul 18. PMID 31219706
- [Result] Duffy AG, Ulahannan SV, Makorova-Rusher O, Rahma O, Wedemeyer H, Pratt D, Davis JL, Hughes MS, Heller T, ElGindi M, Uppala A, Korangy F, Kleiner DE, Figg WD, Venzon D, Steinberg SM, Venkatesan AM, Krishnasamy V, Abi-Jaoudeh N, Levy E, Wood BJ, Greten TF. Tremelimumab in combination with ablation in patients with advanced hepatocellular carcinoma. J Hepatol. 2017 Mar;66(3):545-551. doi: 10.1016/j.jhep.2016.10.029. Epub 2016 Nov 2. PMID 27816492
- [Result] Yau T, Kang YK, Kim TY, El-Khoueiry AB, Santoro A, Sangro B, Melero I, Kudo M, Hou MM, Matilla A, Tovoli F, Knox JJ, Ruth He A, El-Rayes BF, Acosta-Rivera M, Lim HY, Neely J, Shen Y, Wisniewski T, Anderson J, Hsu C. Efficacy and Safety of Nivolumab Plus Ipilimumab in Patients With Advanced Hepatocellular Carcinoma Previously Treated With Sorafenib: The CheckMate 040 Randomized Clinical Trial. JAMA Oncol. 2020 Nov 1;6(11):e204564. doi: 10.1001/jamaoncol.2020.4564. Epub 2020 Nov 12. PMID 33001135
- [Result] Zhu AX, Finn RS, Edeline J, Cattan S, Ogasawara S, Palmer D, Verslype C, Zagonel V, Fartoux L, Vogel A, Sarker D, Verset G, Chan SL, Knox J, Daniele B, Webber AL, Ebbinghaus SW, Ma J, Siegel AB, Cheng AL, Kudo M; KEYNOTE-224 investigators. Pembrolizumab in patients with advanced hepatocellular carcinoma previously treated with sorafenib (KEYNOTE-224): a non-randomised, open-label phase 2 trial. Lancet Oncol. 2018 Jul;19(7):940-952. doi: 10.1016/S1470-2045(18)30351-6. Epub 2018 Jun 3. PMID 29875066
- [Result] Li Z, Liu J, Zhang B, Yue J, Shi X, Cui K, Liu Z, Chang Z, Sun Z, Li M, Yang Y, Ma Z, Li L, Zhang C, Sun P, Zhong J, Zhao L. Neoadjuvant tislelizumab plus stereotactic body radiotherapy and adjuvant tislelizumab in early-stage resectable hepatocellular carcinoma: the Notable-HCC phase 1b trial. Nat Commun. 2024 Apr 16;15(1):3260. doi: 10.1038/s41467-024-47420-3. PMID 38627377
- [Result] Finn RS, Qin S, Ikeda M, Galle PR, Ducreux M, Kim TY, Kudo M, Breder V, Merle P, Kaseb AO, Li D, Verret W, Xu DZ, Hernandez S, Liu J, Huang C, Mulla S, Wang Y, Lim HY, Zhu AX, Cheng AL; IMbrave150 Investigators. Atezolizumab plus Bevacizumab in Unresectable Hepatocellular Carcinoma. N Engl J Med. 2020 May 14;382(20):1894-1905. doi: 10.1056/NEJMoa1915745. PMID 32402160
- [Result] Juloori A, Katipally RR, Lemons JM, Singh AK, Iyer R, Robbins JR, George B, Hall WA, Pitroda SP, Arif F, Fung J, Pillai A, Liao CY, Sharma M, Liauw SL. Phase 1 Randomized Trial of Stereotactic Body Radiation Therapy Followed by Nivolumab plus Ipilimumab or Nivolumab Alone in Advanced/Unresectable Hepatocellular Carcinoma. Int J Radiat Oncol Biol Phys. 2023 Jan 1;115(1):202-213. doi: 10.1016/j.ijrobp.2022.09.052. Epub 2022 Sep 13. PMID 36108891
- [Result] Luke JJ, Onderdonk BE, Bhave SR, Karrison T, Lemons JM, Chang P, Zha Y, Carll T, Krausz T, Huang L, Martinez C, Janisch LA, Hseu RD, Moroney JW, Patel JD, Khodarev NN, Salama JK, Ott PA, Fleming GF, Gajewski TF, Weichselbaum RR, Pitroda SP, Chmura SJ. Improved Survival Associated with Local Tumor Response Following Multisite Radiotherapy and Pembrolizumab: Secondary Analysis of a Phase I Trial. Clin Cancer Res. 2020 Dec 15;26(24):6437-6444. doi: 10.1158/1078-0432.CCR-20-1790. Epub 2020 Oct 7. PMID 33028595
- [Result] Luke JJ, Lemons JM, Karrison TG, Pitroda SP, Melotek JM, Zha Y, Al-Hallaq HA, Arina A, Khodarev NN, Janisch L, Chang P, Patel JD, Fleming GF, Moroney J, Sharma MR, White JR, Ratain MJ, Gajewski TF, Weichselbaum RR, Chmura SJ. Safety and Clinical Activity of Pembrolizumab and Multisite Stereotactic Body Radiotherapy in Patients With Advanced Solid Tumors. J Clin Oncol. 2018 Jun 1;36(16):1611-1618. doi: 10.1200/JCO.2017.76.2229. Epub 2018 Feb 13. PMID 29437535
- [Result] Korpics MC, Polley MY, Bhave SR, Redler G, Pitroda SP, Luke JJ, Chmura SJ. A Validated T Cell Radiomics Score Is Associated With Clinical Outcomes Following Multisite SBRT and Pembrolizumab. Int J Radiat Oncol Biol Phys. 2020 Sep 1;108(1):189-195. doi: 10.1016/j.ijrobp.2020.06.026. Epub 2020 Jun 20. PMID 32569799
- [Result] Onderdonk BE, Chmura SJ. The Yin and Yang of Cytoreductive SBRT in Oligometastases and Beyond. Front Oncol. 2019 Aug 2;9:706. doi: 10.3389/fonc.2019.00706. eCollection 2019. PMID 31428580
- [Result] Dawson LA, Winter KA, Knox JJ, Zhu AX, Krishnan S, Guha C, Kachnic LA, Gillin MT, Hong TS, Craig TD, Williams TM, Hosni A, Chen E, Noonan AM, Koay EJ, Sinha R, Lock MI, Ohri N, Dorth JA, Delouya G, Swaminath A, Moughan J, Crane CH. Stereotactic Body Radiotherapy vs Sorafenib Alone in Hepatocellular Carcinoma: The NRG Oncology/RTOG 1112 Phase 3 Randomized Clinical Trial. JAMA Oncol. 2025 Feb 1;11(2):136-144. doi: 10.1001/jamaoncol.2024.5403. PMID 39699905
- [Result] Abou-Alfa GK, Lau G, Kudo M, Chan SL, Kelley RK, Furuse J, Sukeepaisarnjaroen W, Kang YK, Van Dao T, De Toni EN, Rimassa L, Breder V, Vasilyev A, Heurgue A, Tam VC, Mody K, Thungappa SC, Ostapenko Y, Yau T, Azevedo S, Varela M, Cheng AL, Qin S, Galle PR, Ali S, Marcovitz M, Makowsky M, He P, Kurland JF, Negro A, Sangro B. Tremelimumab plus Durvalumab in Unresectable Hepatocellular Carcinoma. NEJM Evid. 2022 Aug;1(8):EVIDoa2100070. doi: 10.1056/EVIDoa2100070. Epub 2022 Jun 6. PMID 38319892
- [Result] Guo A, Pomenti S, Wattacheril J. Health Disparities in Screening, Diagnosis, and Treatment of Hepatocellular Carcinoma. Clin Liver Dis (Hoboken). 2021 Jun 4;17(5):353-358. doi: 10.1002/cld.1057. eCollection 2021 May. No abstract available. PMID 34136141
- [Result] Yang JD, Hainaut P, Gores GJ, Amadou A, Plymoth A, Roberts LR. A global view of hepatocellular carcinoma: trends, risk, prevention and management. Nat Rev Gastroenterol Hepatol. 2019 Oct;16(10):589-604. doi: 10.1038/s41575-019-0186-y. Epub 2019 Aug 22. PMID 31439937
- See also: Hawai'i Tumor Registry: Cancer at a Glance 2014-2018, a summary of statewide cancer incidence and mortality data used to support regional relevance of the study. — https://www.uhcancercenter.org/research/hawaii-cancer-statistics